CLINICAL TRIAL: NCT05252312
Title: Perception of Nonverbal Acoustic Signals and Resulting Physiological Responses SINOVE-PER
Brief Title: Perception of Nonverbal Acoustic Signals and Resulting Physiological Responses (SINOVE-PER)
Acronym: SINOVE-PER
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University of Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH151; 2020-A02993-36 (Other: ANSM)
Record Dates: First submitted 2022-02-02; First posted 2022-02-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Self Perception
Keywords: nonverbal signals of the vocalizer; nonlinguistic acoustic parameters; physiological responses; perceptual responses; behavioural responses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adult population aged 18 to 80 years: After listening to acoustic stimuli, participants will be asked to judge these stimuli on relevant evaluation criteria (e.g., "how distressed does this person sound?").
  Interventions: Behavioral: Psycho-acoustic tests

INTERVENTIONS:
Behavioral: Psycho-acoustic tests — Listeners' cognitive and biological responses to vocal stimuli will be tested using psycho-acoustic tests. After listening to acoustic stimuli, participants will be asked to judge these stimuli on relevant evaluation criteria (e.g., "how distressed does this person sound?").
  These stimuli might be human voices, animal voices or synthetic voices Physiological measures will be simultaneously taken using an array of complimentary, non-invasive techniques such as the Nociception Level (NOL) Index or video pupillometry

SUMMARY:
Like many other animals, humans produce nonverbal signals including screams, grunts, roars, cries and laughter across a variety of contexts.Due to their acoustic structure, nonverbal vocalizations and valanced speech (e.g., yelling) are also likely to elicit predictable physiological, perceptual or behavioural responses in the receiver of the signal (the listener). This is critical if researchers are to gain a comprehensive understanding of the broad range of mechanisms and the evolved functions of acoustic communication.

Therefore, in this research, investigators will examine specifically how exposure to vocal stimuli affects both the cognitive and biological responses of the listener.

DETAILED DESCRIPTION:
Like many other animals, humans produce nonverbal signals including screams, grunts, roars, cries and laughter across a variety of contexts. Many of these signals (such as cries) are already produced at birth and are likely to serve a number of important biological and social functions. In addition, human speech is characterized by nonlinguistic acoustic parameters (such as pitch, formant frequencies, and nonlinear phenomena) that are known to correlate with biologically important traits of the vocalizer.

Due to their acoustic structure, nonverbal vocalizations and valanced speech (e.g., yelling) are also likely to elicit predictable physiological, perceptual or behavioural responses in the receiver of the signal (the listener).

However, while a number of playback studies have examined behavioural responses (e.g., ratings) of listeners when exposed to various voice stimuli, very few studies have examined whether such behavioural responses are accompanied by an underlying physiological response. This is critical if researchers are to gain a comprehensive understanding of the broad range of mechanisms and the evolved functions of acoustic communication.

Therefore, in this research, investigators will examine specifically how exposure to vocal stimuli affects both the cognitive and biological responses of the listener.

ELIGIBILITY:
Inclusion Criteria:

- Participant should be affiliated or entitled to a social security scheme

Exclusion Criteria:

* Pregnancy
* Hearing impairment, speech production disorders or major health problems.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult population aged 18 to 80 years
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of correct responses in a forced-choice task after vocal stimuli | Immediately after the vocal stimuli
  Participants will be asked to judge vocal stimuli Example : "Of the two baby cries you listened to, which one do you think shows the most distress"
Numerical values of judgements along a scale | Immediately after the vocal stimuli
  Participants will be asked to judge vocal stimuli Example : participants may be asked to judge, along a gradient (from 0 to 100), "how consistent the distress of the baby you heard is to you".
Response time (second) | Immediately after the vocal stimuli
  Participants will be asked to judge vocal stimuli In this case, the participant is instructed to respond as soon as possible. The response time for each stimulus is then systematically measured

SECONDARY OUTCOMES:
Heart rate (bpm) | During the vocal stimuli
Skin conductance (Siemens) | During the vocal stimuli
Skin temperature (°C) | During the vocal stimuli
Nociception Level Index (NOL) | During the vocal stimuli
  A non-invasive finger probe, containing four sensors, will be placed on the on the index finger of the participants.
Pupillary diameter (millimeter) | During the vocal stimuli
  Using a high resolution binocular for automated pupil diameter measurement with an infrared camera

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND PEYRON, MDPHD, Principal Investigator — CHU DE SAINT-ETIENNE; Nicolas MATHEVON, PhD, Study Chair — University of Saint-Etienne, France
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No